CLINICAL TRIAL: NCT00025363
Title: A Groupwide Randomized Phase II Window Study of Two Different Schedules of Irinotecan in Combination With Vincristine And Pilot Assessment of Safety and Efficacy of Tirapazamine Combined With Multiagent Chemotherapy for First Relapse or Progressive Disease in Rhabdomyosarcoma and Related Tumors
Brief Title: Comparison of Chemotherapy Regimens in Treating Children With Relapsed or Progressive Rhabdomyosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01864; ARST0121; U10CA098543 (NIH); CDR0000068954 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Alveolar Childhood Rhabdomyosarcoma; Embryonal Childhood Rhabdomyosarcoma; Embryonal-botryoid Childhood Rhabdomyosarcoma; Previously Treated Childhood Rhabdomyosarcoma; Recurrent Childhood Rhabdomyosarcoma
MeSH Terms: interventions — Vincristine; Irinotecan; Cyclophosphamide; Doxorubicin; Ifosfamide; indolepropanol phosphate; Etoposide; Tirapazamine; Filgrastim; Granulocyte Colony-Stimulating Factor; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Pharmacogenomic Testing

ARMS (2):
- Arm I (Experimental): Patients receive vincristine IV on days 1 and 8 and irinotecan IV over 1 hour on days 1-5 and 8-12. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vincristine sulfate; Drug: irinotecan hydrochloride; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: ifosfamide; Drug: etoposide; Drug: tirapazamine; Biological: filgrastim; Biological: sargramostim; Other: pharmacological study; Other: pharmacogenomic studies; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients receive vincristine IV on days 1 and 8 and irinotecan IV over 1 hour on days 1-5. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vincristine sulfate; Drug: irinotecan hydrochloride; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: ifosfamide; Drug: etoposide; Drug: tirapazamine; Biological: filgrastim; Biological: sargramostim; Other: pharmacological study; Other: pharmacogenomic studies; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: ifosfamide — Given IV
  Other Names: Cyfos; Holoxan; IFF; IFX; IPP
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: tirapazamine — Given IV
  Other Names: SR 4233; Tirazone; WIN 59075
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Biological: sargramostim — Given SC
  Other Names: GM-CSF; Leukine; Prokine
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: pharmacogenomic studies — Correlative studies
  Other Names: Pharmacogenomic Study
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Randomized phase II trial to compare the effectiveness of different combination chemotherapy regimens in treating children who have rhabdomyosarcoma. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare response rate in children with relapsed or progressive rhabdomyosarcoma, undifferentiated sarcoma, or ectomesenchymoma treated with 2 different schedules of irinotecan and vincristine in an upfront phase II window.

II. Determine the progression-free and overall survival of patients treated with multiagent chemotherapy.

III. Determine the toxic effects of tirapazamine, doxorubicin, and cyclophosphamide in these patients.

IV. Determine the toxic effects of irinotecan and vincristine in these patients.

V. Determine whether conversion of irinotecan to its active metabolite SN-38 predicts tumor response in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to risk status and window therapy eligibility (unfavorable risk and eligible vs unfavorable risk and ineligible vs favorable risk).

UNFAVORABLE-RISK PATIENTS ELIGIBLE FOR WINDOW THERAPY: Patients are stratified according to prior topotecan (yes vs no). These patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive vincristine IV on days 1 and 8 and irinotecan IV over 1 hour on days 1-5 and 8-12. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive vincristine IV on days 1 and 8 and irinotecan IV over 1 hour on days 1-5. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

Patients in both arms with partial response (PR) or complete response (CR) receive 5 additional courses of irinotecan and vincristine on the previous schedule. In addition, patients with PR or CR also receive cyclophosphamide/doxorubicin (CD) and ifosfamide/etoposide (IE) chemotherapy.

CD/IE CHEMOTHERAPY: Patients receive cyclophosphamide IV over 1 hour and doxorubicin IV over 15-30 minutes on day 1 of weeks 7, 16, 28, 37, and 40. Patients also receive ifosfamide IV over 1 hour and etoposide IV over 1 hour on days 1-5 of weeks 10, 19, 22, 31, and 43. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients with no response or progressive disease on arm I or II proceed to tirapazamine/cyclophosphamide/doxorubicin (TCD) and ifosfamide/etoposide (IE) chemotherapy.

TCD/IE CHEMOTHERAPY: Patients receive tirapazamine IV over 2 hours, cyclophosphamide IV over 1 hour, and doxorubicin IV over 15-30 minutes on day 1 of weeks 7, 10, 16, 25, and 34. Patients also receive ifosfamide IV over 1 hour and etoposide IV over 1 hour on days 1-5 of weeks 13, 19, 22, 28, 31, and 37.

PATIENTS WITH UNFAVORABLE RISK AND INELIGIBLE FOR WINDOW THERAPY: Patients receive tirapazamine IV over 2 hours, cyclophosphamide IV over 1 hour, and doxorubicin IV over 15-30 minutes on day 1 of weeks 1, 4, 10, 19, and 28. Patients also receive ifosfamide IV over 1 hour and etoposide IV over 1 hour on days 1-5 of weeks 7, 13, 16, 22, 25, and 31. Patients also receive filgrastim (G-CSF) or sargramostim (GM-CSF) subcutaneously (SC) beginning 1 day after each course of chemotherapy and continuing until blood counts recover. Treatment continues in the absence of disease progression or unacceptable toxicity.

PATIENTS WITH FAVORABLE RISK: Patients receive cyclophosphamide IV over 1 hour and doxorubicin IV over 15-30 minutes on day 1 of weeks 1, 4, 10, 19, and 28. Patients also receive ifosfamide IV over 1 hour and etoposide IV over 1 hour on days 1-5 of weeks 7, 13, 16, 22, 25, and 31. Patients also receive G-CSF or GM-CSF SC beginning 1 day after each course of chemotherapy and continuing until blood counts recover. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 1 year, every 4 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rhabdomyosarcoma, undifferentiated sarcoma, or ectomesenchymoma

  * First relapse or first occurrence of disease progression
* Unfavorable-risk patients eligible for study window therapy with irinotecan and vincristine meeting the following criteria:

  * Unfavorable risk defined by any of the following:

    * Embryonal histology with stage I or group I at initial diagnosis with distant recurrence or with local or regional recurrence after prior cyclophosphamide
    * Embryonal histology with initial stage II, III, or IV or group II, III, or IV with any relapse pattern
    * Alveolar histology with any stage or group at initial diagnosis
  * At least unidimensionally measurable disease
  * No prior irinotecan
  * Bone marrow must not be only site of relapse
* Unfavorable-risk patients ineligible for study window therapy with irinotecan meeting the following criteria:

  * Either no measurable disease OR patient received prior irinotecan
  * Bone marrow as only site of relapse allowed
* Favorable-risk patients meeting the following criteria:

  * Initial botryoid histology (any stage, any group, or any pattern of relapse)
  * Embryonal histology if either stage I or group I (with either local or regional recurrence)
  * No prior cyclophosphamide
* No CNS metastases
* Performance status - ECOG 0-2
* Performance status - Zubrod 0-2
* At least 2 months
* Absolute neutrophil count at least 750/mm^3
* Platelet count at least 75,000/mm^3 (transfusion independent)
* Hemoglobin at least 10.0 g/dL (red blood cell transfusion allowed)
* Bilirubin no greater than 1.5 times normal
* SGPT less than 2.5 times normal
* Creatinine no greater than 1.5 times normal
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min
* Shortening fraction at least 27% by echocardiogram
* Ejection fraction at least 50% by MUGA
* No prior ischemic heart disease
* Seizure disorder allowed if well controlled by anticonvulsants
* No CNS toxicity greater than grade 2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior myeloablative therapy with stem cell transplantation
* At least 1 week since prior antineoplastic biologic agent
* At least 1 week since prior growth factor(s)
* Recovered from prior immunotherapy
* No concurrent immunomodulating agents
* See Disease Characteristics
* See Biologic therapy
* No more than 1 prior chemotherapy regimen
* No prior doxorubicin or daunorubicin
* At least 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No other concurrent anticancer chemotherapy
* Concurrent corticosteroid therapy allowed
* At least 2 weeks since prior small-port radiotherapy.
* At least 6 months since prior radiotherapy to 50% or more of pelvis
* At least 6 weeks since other prior substantial radiotherapy to bone marrow
* Recovered from prior radiotherapy
* Concurrent radiotherapy to localized painful lesions allowed provided at least 1 measurable lesion is not irradiated
* No concurrent intensity-modulated radiotherapy

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2001-11; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Response at week 6 of investigational window therapy (unfavorable risk patients) | At week 6
Incidence of DLT when tirapazamine is given in combination with cyclophosphamide and doxorubicin, graded according to the NCI CTC v 2.0 | Up to 6 years

SECONDARY OUTCOMES:
Incidence of toxicities associated with the two administration schedules of irinotecan in combination with vincristine, graded according to the NCI CTC v 2.0 (unfavorable risk patients) | Up to 6 years
Blood metabolite SN-38 levels (unfavorable risk patients) | Up to 6 years
Progression-free survival | Up to 6 years
Survival | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Philip Breitfeld, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States